CLINICAL TRIAL: NCT07048652
Title: Evaluating the Diagnostic Performance of High-Resolution Computed Tomography (HRCT) in Detecting Idiopathic Pulmonary Fibrosis (IPF) in Suspected Cases
Brief Title: Evaluating the Diagnostic Performance of (HRCT) in IPD Fibrosis in Suspected Cases
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/905
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High-Resolution Computed Tomography — High-resolution computed tomography (HRCT) plays a crucial role in diagnosing and managing Idiopathic Pulmonary Fibrosis (IPF). It helps identify the characteristic pattern of IPF, known as Usual Interstitial Pneumonia (UIP), and can sometimes obviate the need for lung biopsy.

SUMMARY:
This will be a cross-sectional descriptive study aimed at evaluating the role of high-resolution computed tomography (HRCT) in diagnosing Idiopathic Pulmonary Fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above.
* Patients clinically suspected of having IPF.
* Patients referred for HRCT examination.
* Patients who provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with a known diagnosis of other interstitial lung diseases.
* Patients with comorbid conditions that could mimic IPF.
* Patients who are pregnant.
* Patients with incomplete medical records or imaging studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic Pulmonary Fibrosis (IPF): IPF is defined as a chronic, progressive fibrotic interstitial lung disease diagnosed based on clinical evaluation, exclusion of other potential causes, and characteristic radiological findings on high-resolution CT (HRCT).
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
high-resolution computed tomography (HRCT) | 12 Months
  Idiopathic Pulmonary Fibrosis (IPF) high-resolution computed tomography (HRCT) scans are crucial for diagnosis and assessment of disease severity. HRCT findings typically show a reticular pattern with traction bronchiectasis and honeycombing, predominantly in the subpleural and basal regions of the lungs

CONTACTS AND LOCATIONS:
Locations (1):
- AYK Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No